CLINICAL TRIAL: NCT03779139
Title: A Randomized Trial of Intra-Portal Alone Versus Intra- and Extra-Portal Transplantation of Pancreatic Islets After Total Pancreatectomy for Chronic Pancreatitis
Brief Title: Intra-Portal Alone Versus Intra- and Extra-Portal Transplantation of Pancreatic Islets After Total Pancreatectomy for Chronic Pancreatitis
Acronym: iSite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURG-2017-26057
Record Dates: First submitted 2018-11-05; First posted 2018-12-19 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pancreatitis; Diabetes Mellitus; Islet Cell Transplantation
Keywords: total pancreatectomy with islet autotransplant
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrahepatic islets alone (Active Comparator)
  Interventions: Procedure: Intrahepatic islets alone
- Intrahepatic and omental pouch islets (Experimental)
  Interventions: Procedure: Intrahepatic islets and islets in the omental pouch
- Normal Volunteers (Sham Comparator)
  Interventions: Other: Normal Volunteers

INTERVENTIONS:
Procedure: Intrahepatic islets and islets in the omental pouch — Patients with islet harvest of >5000 islet equivalents per kg body weight will be randomized in a 1:1 ratio to 4000 IEq/kg delivered via intraportal route and the remainder implanted into a constructed omental pouch.
  Arms: Intrahepatic and omental pouch islets
Procedure: Intrahepatic islets alone — This is the standard of care procedure. Patients with islet harvest of >5000 islet equivalents per kg body weight will be randomized in a 1:1 ratio to all islets autotransplanted intrahepatically via the intraportal route.
  Arms: Intrahepatic islets alone
Other: Normal Volunteers — These individuals will undergo metabolic testing as well as islet cell function testing.
  Arms: Normal Volunteers

SUMMARY:
Randomized pilot trial of patients (n=30) undergoing Total Pancreatectomy and Islet AutoTransplant (TPIAT). Patients with islet harvest of greater than 5000 islet equivalents/kg body weight will be randomized to receive a portion of their islets into an omental pouch. For outcomes related to islet function, a group of normal volunteers (n=15) will be studied as a comparator group.

DETAILED DESCRIPTION:
Chronic pancreatitis affects as many as 1 in every 2,500 persons and is associated with incapacitating pain, frequent hospitalization and risk of narcotic dependence. This is a debilitating disease with limited treatment options; afflicted patients are often young or middle aged adults. The health and economic costs of pancreatitis are great. Nearly $300 million is spent on emergency department visits alone in the US each year. More than 90% of patients with chronic pancreatitis have been hospitalized, half use narcotic analgesics regularly, and one-fourth are on disability. The lifetime risk of diabetes mellitus is as high as 70%. This proposal addresses needs in two broad topic areas: pancreatitis, and diabetes. The investigators propose to investigate a new technique for implanting autologous pancreatic islet cells into patients undergoing surgery for acute recurrent or chronic pancreatitis in an effort to improve long-term diabetes control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-68
2. Scheduled for total pancreatectomy and IAT at U of MN. All patients who are approved for pancreatectomy and IAT at U of MN are reviewed by a multi-disciplinary committee including surgeons, gastroenterologists specializing in pancreatic disease, a pain specialist psychologist, and endocrinologist to confirm the diagnosis of chronic pancreatitis and candidate suitability for surgery.
3. Able to provide informed consent

Exclusion Criteria:

1. Pre-Existing diabetes mellitus fasting blood glucose>115mg/dl, or hemoglobin A1c level >6.0% because these are all evidence of inadequate beta-cello mass.
2. Use of any of the following treatments in the 30 days prior to enrollment: insulin, metformin, sulfonylureas, glinides, thiazolidinediones, GLP-1 agonists, DPP-4 inhibitors, or amylin.
3. ALT or AST>2.5 times the upper limit of normal (ULN). Bilirubin>ULN, unless due to benign diagnosis such as Gilbert's.
4. Any of the following hematologic abnormalities: server anemia (hemoglobin <10 g/dL), thrombocytopenia (<150/mm3), or neutropenia(<1.0 x 109/L).
5. Current use or expected use of oral or injected corticosteroids, or any mediation likely to affect glucose tolerance. However, use of hydrocortisone for physiologic replacement, or use of any topical, inhaled or intranasal glucocorticoid is permitted.
6. Current or expected use of any other immunosuppressive agent.
7. Known coagulopathy, or need for anticoagulant therapy preoperatively (coumadin, enoxaparin), or any history of pulmonary embolism.
8. For females, plans to become pregnant or unwillingness to use birth control for the study duration.
9. Inability to comply with the study protocol.
10. Untreated psychiatric illness that may interfere with ability to give informed consent, or other developmental delay or neurocognitive disorder that impairs with a patient's ability to consent on their own behalf.
11. Any other medical condition that , in the opinion of the investigator, may interfere wit the patient's ability to successfully and safely complete the trial.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Portal vein thrombosis | Post operative day 4 or 5.
  Portal vein thrombosis is associated with higher tissue volume infused into the portal vein and higher portal pressures and is assessed using abdominal ultrasound.
Clavien-Dindo classification of surgical complications | Within 30 days of surgery
  Grades surgical complications based on the level of treatment necessary to treat the complication.
Mixed Meal Tolerance Test | 1 year
  Patient is given Boost HP (6cc/kg), ingested 5 minutes after t=0 blood draw. Blood is drawn every half hour for 2 hours.
Intravenous Glucose tolerance test | 1 year
  Patients are given a bolus of 0.2mg/kg of dextrose at t=0. Blood samples will be drawn at t=-10,-5,-1,2,3,4,5,7 and 10 minutes
Glucose potentiated arginine stimulation | 1 year
  Starting immediately after glucose tolerance test (time t=10 minutes), 20% dextrose will be infused to maintain a glucose ~230mg/dL until test is completed. Glucose levels are measured every 5 minutes to maintain glucose in the target range after 40 minutes of continuous 20% dextrose infusion, After 40 minutes of continuous D20% infusion, baseline samples for glucose, insulin, and C-peptide are drawn (three samples over 10 minutes), a bolus of 5 grams arginine is given (at time 55 minutes), and samples for glucose, insulin, and C-peptide are taken at 2, 3, 4, and 5 minutes after
  the arginine bolus.
Hypoglycemic clamp | 1 year
  A stepped hypoglycemic clamp protocol with variable glucose infusion rates will be performed to achieve 45 min glucose plateaus at 70, 60, and 50 mg/dl.Glucagon responses will be calculated by subtracting the mean of the three baseline values observed prior to the clamp from glucagon levels observed at 70, 60, and 50 mg/dl glucose nadirs during the clamp
Continuous glucose monitoring | 1 year
  3 days of CGM monitoring at one year will be obtained for mean glucose,standard deviation, and percent of time in hypo- and hyperglycemia
Hemoglobin A1c levels | 1 year
  Measure of average glucose levels over last several weeks
Insulin Use | 1 year
  calculated as units/kg/day, will be assessed from glucose and insulin diaries maintained by patients for 14 days, overlapping with day 90
Hypoglycemic episodes | 1 year
  All severe hypoglycemic events will be recorded. This is defined based on American Diabetes Association criteria as a hypoglycemic episode <54 mg/dL or (if not measured) associated with prompt recovery upon administration of glucose in which a patient is mentally or physically incapacitated and requires assistance from another person to treat the hypoglycemia.
Clarke score | 1 year
  is determined from eight questions characterizing the participant's exposure to episodes of moderate and severe hypoglycemia; it evaluates symptomatic responses to hypoglycemia. A score of 4 or greater suggests impaired awareness of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Greg Beilman, MD, Principal Investigator — University of Minnesota, Department of Surgery
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No